CLINICAL TRIAL: NCT00376675
Title: Long Acting Methylphenidate (Concerta™) for Cancer-Related Fatigue: A Phase III, Randomized, Double-Blind Placebo Controlled Study
Brief Title: Methylphenidate in Treating Patients With Fatigue Caused by Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N05C7; NCI-2012-02701 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000495148 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Results first posted 2014-10-10 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Fatigue; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: fatigue; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Fatigue | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral methylphenidate hydrochloride daily on days 1-28.
  Interventions: Drug: methylphenidate hydrochloride
- Arm II (Placebo Comparator): Patients receive oral placebo daily on days 1-28.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: methylphenidate hydrochloride — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Methylphenidate may help relieve fatigue caused by cancer. It is not yet known whether methylphenidate is more effective than a placebo in relieving fatigue and improving quality of life in patients with cancer.

PURPOSE: This randomized phase III trial is studying methylphenidate to see how well it works in treating patients with fatigue caused by cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Test the efficacy of long-acting methylphenidate in patients with cancer-related fatigue as measured using an item of the Brief Fatigue Inventory.

Secondary

* Evaluate the tolerability and adverse events associated with this drug in these patients.
* Study the effect of this drug on quality of life (QOL)-related variables (vitality, sleep quality, overall QOL, QOL domains, other fatigue measures, and perceived treatment efficacy) in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to disease stage (0, I, or II vs III or IV), level of fatigue at baseline (4-7 vs 8-10), concurrent biological therapy (yes vs no), concurrent chemotherapy (yes vs no), and concurrent radiotherapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral methylphenidate daily on days 1-28.
* Arm II: Patients receive oral placebo daily on days 1-28.

Patients in both arms complete questionnaires to assess their symptoms of fatigue, overall mood, quality of life, sleep quality, and adverse effects from treatment at baseline and once weekly for 4 weeks. Patients also complete a Symptom Experience Diary.

McNeil Consumer & Specialty Pharmaceuticals provided medication support for NCCTG N05C7.

PROJECTED ACCRUAL: A total of 140 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Men or women with a history of cancer-related fatigue as defined by a score ≥ 4 on a fatigue numerical analogue scale (0 - 10)
3. Fatigue for ≥ 1 month prior to registration
4. ECOG Performance Score (PS) 0, 1, or 2
5. Life expectancy ≥ 6 months
6. Histologic or cytologic proven cancer other than brain cancer or CNS lymphoma
7. Laboratory values obtained ≤ 30 days prior to registration:

   * Hgb ≥ 10 g/dL
8. Willing and able to provide informed consent
9. Negative pregnancy test (urine or serum) done ≤ 7 days prior to registration, for women of childbearing potential only
10. Ability to complete questionnaire(s) by themselves or with assistance
11. Biological therapy (i.e. immunotherapy, biotherapy), chemotherapy or radiation therapy will be allowed
12. Use of a stable dose of anti-depressants (except tricyclic anti-depressants) will be allowed
13. Erythropoietic agents to treat anemia, and steroids as a part of cancer treatment and for symptom management (except for fatigue) will be allowed

Exclusion Criteria:

1. Hypersensitivity to methylphenidate
2. Any prior use of methylphenidate
3. Concomitant (≤ 2 weeks) use of prescription stimulants (pemoline, modafinil, amphetamines); other medications, herbal products or dietary supplements for fatigue
4. Uncontrolled hypertension [defined as systolic blood pressure (BP) ≥ 160 mmHg and/or diastolic BP ≥ 100 mmHg on 2 separate visits ≤ 2 months prior to randomization]; or a resting heart rate > 100
5. Moderate or severe pain as defined by an average daily score ≥ 4 on a pain analog scale (0 - 10)
6. Known brain metastasis or primary CNS malignancy
7. Clinically significant acute or chronic progressive or unstable neurologic (dementia, delirium, or seizure disorder), hepatic, renal, cardiovascular, thyroid, or respiratory disease that would limit participation in the study per MD discretion or judgment
8. Psychiatric disorder such as manic depression, anxiety disorder, bipolar disorder, obsessive compulsive disorder, or schizophrenia
9. Major surgery < 4 weeks prior to registration. (Note: Insertion of central venous catheter is not considered major surgery.)
10. Using a drug contraindicated when taken concurrently with methylphenidate: coumarin anticoagulants, anticonvulsants, tricyclic antidepressants, antipsychotics, monoamine oxidase inhibitors, clonidine, theophylline, and pseudoephedrine

    Note: use of Compazine prescribed as an antiemetic is permitted for use while participating in this study.
11. Additional medical conditions where use of methylphenidate is contraindicated:

    glaucoma, motor tics, family history or diagnosis of Tourette's syndrome, history of drug or alcohol abuse or intestinal obstruction.
12. Pregnant women or nursing women. Women of childbearing potential who are unwilling to employ adequate contraception. This study involves an investigational agent whose genotoxic, mutagenic, and teratogenic effects on the developing fetus and newborn are unknown.
13. Untreated hypothyroidism (TSH ≥ 5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2008-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sood, MD, Study Chair — Mayo Clinic
Locations (238):
- United States (238):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Mercy Hospital at Wilkes-Barre, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Southlake Clinic, Renton, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Moraska AR, Sood A, Dakhil SR, Sloan JA, Barton D, Atherton PJ, Suh JJ, Griffin PC, Johnson DB, Ali A, Silberstein PT, Duane SF, Loprinzi CL. Phase III, randomized, double-blind, placebo-controlled study of long-acting methylphenidate for cancer-related fatigue: North Central Cancer Treatment Group NCCTG-N05C7 trial. J Clin Oncol. 2010 Aug 10;28(23):3673-9. doi: 10.1200/JCO.2010.28.1444. Epub 2010 Jul 12. PMID 20625123

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One-hundred and forty-eight (148) participants were recruited between February 2008 and August 2008 from 20 North Central Treatment Group (NCCTG) member sites.
Pre-assignment Details: There were a total of 8 cancellations (5 Methylphenidate, 3 Placebo) and 1 ineligible participant on Placebo. These 9 participants were excluded from all analysis.
Groups:
- Methylphenidate: Patients receive oral methylphenidate daily on days 1-28.
- Placebo: Patients receive oral placebo daily on days 1-28.
Period: Overall Study
Arm/Group | Methylphenidate | Placebo
Started | 69 | 70
Completed | 49 | 56
Not Completed | 20 | 14
Not completed — Withdrawal by Subject | 9 | 2
Not completed — Adverse Event | 10 | 5
Not completed — Other Reason | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate | Placebo | Total
Number analyzed (Participants) | 69 | 70 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (11.23) | 60.6 (13.82) | 59.9 (12.58)
Age, Customized [Number; unit: participants]
  <50 years | 14 | 14 | 28
  >=50 years | 55 | 56 | 111
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 40 | 84
  Male | 25 | 30 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 66 | 64 | 130
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 69 | 70 | 139
Current chemotherapy [Number; unit: participants]
  Yes | 44 | 45 | 89
  No | 25 | 25 | 50
Curative intent treatment [Number; unit: participants]
  Missing | 0 | 2 | 2
  Yes | 34 | 30 | 64
  No | 35 | 38 | 73
Concurrent radiation [Number; unit: participants]
  Yes | 9 | 7 | 16
  No | 60 | 63 | 123
Concurrent biological therapy [Number; unit: participants]
  Yes | 17 | 17 | 34
  No | 52 | 53 | 105
Fatigue scale [Number; unit: participants] — Fatigue was measured using a scale of 0 to 10, with 0 (No fatigue) and 10 (Fatigue as bad as you can imagine).
  participants
    4-7 | 47 | 48 | 95
    8-10 | 22 | 22 | 44
Stage [Number; unit: participants] — Stage 0: Carcinoma in situ; Stage I, II and III: Higher numbers indicate more extensive disease: larger tumor size and/or spread of the cancer beyond the organ in which it first developed to nearby lymph nodes and/or tissues or organs adjacent to the location of the primary tumor; Stage IV: The cancer has spread to distant tissues or organs
  participants
    0/I/II | 22 | 22 | 44
    III/IV | 47 | 48 | 95
Type of cancer [Number; unit: participants]
  Breast | 26 | 20 | 46
  Colon | 4 | 4 | 8
  Prostate | 2 | 6 | 8
  Lung | 10 | 8 | 18
  Combination/Unknown/Other | 27 | 32 | 59
Average fatigue over the last week [Mean (Standard Deviation); unit: units on a scale] — Fatigue was measured in a scale of 0 to 100 with 0 (poor quality of life or bad symptoms) and 100 (best quality of life or no symptoms).
  units on a scale | 33.6 (15.43) | 34.0 (17.23) | 33.8 (16.30)
Average pain over the last 24 hours [Mean (Standard Deviation); unit: units on a scale] — Pain was measured in a scale of 0 to 100 with 0 (poor quality of life or bad symptoms) and 100 (best quality of life or no symptoms).
  units on a scale | 87 (13.88) | 86 (12.58) | 86.3 (13.20)

OUTCOME MEASURES:

1. Primary Outcome: Prorated AUC of Total Fatigue as Measured by the Brief Fatigue Inventory (BFI) at Baseline and at Weeks 1-4
Description: The prorated area under the curve (AUC) for the usual fatigue question of the BFI at baseline and at weeks 1-4 after being translated onto a 0 (poor quality of life (QOL) or bad symptoms) to 100 (best QOL or no symptoms) point scale was calculated as the following:
  1. For those completed 4 weeks item: AUC/4;
  2. For those completed up to week 3 item: (AUC * 4) / 3;
  3. For those completed up to week 2 item: AUC * 2;
  4. For those completed up to week 1 item: AUC * 4;
  The prorated AUC scores were then transformed onto 0 to 100 point scale with 0 (poor QOL or bad symptoms) and 100 (best QOL or no symptoms) for analysis.
Time Frame: Baseline to week 4
Population: All participants meeting the eligibility criteria who have signed a consent form, started treatment, and provided a baseline and one post-baseline usual fatigue score were evaluable for this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 62 | 63
units on a scale | 50.33 (20.32) | 47.15 (17.00)
Statistical Analysis 1: Comparison: Methylphenidate vs Placebo; Test type: Superiority or Other; p = 0.317, Wilcoxon rank sum test

2. Secondary Outcome: Severity of Adverse Events as Measured by the Symptom Experience Diary Based on Mean Changes From Baseline to Week 4
Description: The Symptom Experience Diary (SED) consists of 12 items. All scores were translated onto a 0-100 point scale, with 0 represent poor quality of life (QOL) or bad symptom and 100 is best QOL or no symptoms.The change in severity of adverse events was calculated as subtracting the item scores at baseline from the scores at week 4.
Time Frame: Baseline and Week 4
Population: All participants who have provided a baseline and week 4 SED scores were evaluable for this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 49 | 56
units on a scale
  Nervousness | -2.7 (20.08) | 9.5 (17.15)
  Appetite decrease | -5.2 (21.04) | 6.6 (28.87)
  Sex drive | -0.9 (22.63) | 9.8 (37.17)
  Abdominal pain | -3.5 (21.85) | 3.6 (19.49)
  Dizziness | -2.2 (15.58) | 2.1 (17.76)
  Shakiness | -0.6 (11.97) | 1.4 (18.82)
  Heartbeat | -2.0 (10.60) | -1.6 (16.60)
  Vomiting | -0.8 (9.19) | 0.4 (18.29)
  Headaches | -0.8 (18.80) | 3.9 (17.34)
  Trouble sleeping | 10.6 (29.99) | 11.1 (28.58)
  Fatigue distress | 22.9 (32.94) | 15.8 (33.25)
  Fatigue control satisfaction | 28.0 (32.77) | 23.2 (34.57)

3. Secondary Outcome: AUC of Sleep Quality as Measured by the Pittsburgh Sleep Quality Index at Baseline and at Weeks 1-4
Description: Pittsburgh Sleep Quality Index (PSQI) consists of 19 items and 7 scales. The AUC for the overall PSQI at baseline and at weeks 1-4 after being translated onto a 0 to 100 point scale was calculated. Higher scores are better.
Time Frame: Baseline to Week 4
Population: All participants who have provided a baseline and one post-baseline PSQI score were evaluable for this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale * weeks
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 63 | 65
units on a scale * weeks | 144.37 (110.32) | 145.93 (108.21)

4. Secondary Outcome: AUC of Vitality as Measured by the Short Form-36 Vitality Subscale at Baseline and at Weeks 1-4
Description: The SF-36 is a 36-item short form to measure health status in various populations. The vitality subscale is comprised of 4 items and is a measure of energy level as well as fatigue. The AUC for the vitality subscale at baseline and at weeks 1-4 after being translated onto a 0 to 100 point scale was calculated. Higher scores are better.
Time Frame: Baseline to Week 4
Population: All participants who have provided a baseline and one post-baseline Vitality subscale score were evaluable for this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale * weeks
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 69 | 68
units on a scale * weeks | 134.74 (88.77) | 121.59 (76.31)

5. Secondary Outcome: AUC of Overall Quality of Life (QOL) and QOL Domains as Measured by the Linear Analogue Self Assessment at Baseline and at Weeks 1-4
Description: Linear Analogue Self Assessment (LASA) consists of 6 single-item numeric analogue scales. The AUC for the six-items at baseline and at weeks 1-4 after being translated onto a 0 to 100 point scale was calculated. Higher scores are better.
Time Frame: Baseline to Week 4
Population: All participants who have provided a baseline and one post-baseline LASA score were evaluable for this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale * weeks
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 68 | 68
units on a scale * weeks
  Overall QOL | 204.21 (103.16) | 201.34 (94.65)
  Mental well-being | 227.04 (109.61) | 226.40 (100.62)
  Physical well-being | 188.13 (98.12) | 191.07 (87.23)
  Emotional well-being | 203.65 (105.32) | 215.65 (96.90)
  Social activity | 189.68 (112.89) | 177.34 (95.99)
  Spiritual well-being | 231.24 (122.30) | 255.88 (113.74)

6. Secondary Outcome: AUC of Other Fatigue Scores as Measured by Items of the Brief Fatigue Inventory (BFI) at Baseline and at Weeks 1-4
Description: Area under the curve (AUC) for the other fatigue items of the BFI at baseline and at weeks 1-4 after being translated onto a 0 to 100 point scale was calculated. Higher scores are better.
Time Frame: Baseline to Week 4
Population: All participants who have provided a baseline and one post-baseline BFI score were evaluable for this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale * weeks
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 68 | 69
units on a scale * weeks
  Fatigue right now | 179.96 (100.06) | 174.94 (92.95)
  Worst fatigue last 24 hours | 144.59 (92.95) | 126.36 (82.13)
  Fatigue interference with general activity | 187.60 (106.88) | 171.06 (98.11)
  Fatigue interference with mood | 205.31 (106.89) | 220.29 (114.85)
  Fatigue interference with walking ability | 210.09 (125.36) | 206.46 (120.76)
  Fatigue interference with normal work | 179.94 (106.40) | 168.84 (104.20)
  Fatigue interference with relations with others | 224.72 (114.46) | 243.87 (115.95)
  Fatigue interference with enjoyment of life | 194.15 (115.11) | 184.12 (111.10)

7. Secondary Outcome: Anchor-based Minimally Important Difference in SGIC Overall Quality of Life Based on Mean Changes From Baseline to Week 4 on BFI Usual Fatigue
Description: Perceived treatment efficacy was measured by the Subject Global Impression of Change (SGIC). The SGIC is a 3-point item in which the patient rates the change in the overall status since beginning the study drug (ranging from very much better, moderately better, a little better, about the same, a little worse, moderately worse, to very much worse). The average change in patient fatigue scores for those participants who express a perceived change of "a little better" via the SGIC scores were calculated. BFI usual fatigue item score was translated into 0 to 100 point scale for the analysis, with 0 (poor QOL or bad symptoms) and 100 (best QOL or no symptoms).
Time Frame: Baseline and Week 4
Population: All participants who have provided a baseline and week 4 BFI usual fatigue scores and a perceived change of "a little better" via SGIC scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 11 | 10
units on a scale | 20.9 (18.1) | 15 (22.2)

8. Secondary Outcome: Anchor-based Minimally Important Difference in SGIC Physical Condition Based on Mean Changes From Baseline to Week 4 on BFI Usual Fatigue
Description: as for outcome 7
Time Frame: Baseline and Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 13 | 7
Units on scale | 20.0 (14.7) | 11.4 (27.3)

9. Secondary Outcome: Anchor-based Minimally Important Difference in SGIC Emotional State Based on Mean Changes From Baseline to Week 4 on BFI Usual Fatigue
Description: as for outcome 7
Time Frame: Baseline and Week 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 10 | 13
Units on scale | 31.0 (24.7) | 23.8 (29.3)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: One participant on Methylphenidate and one participant on placebo did not have adverse event data provided post baseline.
Arm/Group | Methylphenidate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/69
Other Adverse Events (participants affected / at risk) | 56/68 | 54/69
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methylphenidate (N=68) | Placebo (N=69)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 16 (33) | 21 (53)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Disease progression (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (5) | 4 (9)
Fever (General disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (3)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Dizziness (Nervous system disorders) | 18 (40) | 25 (58)
Headache (Nervous system disorders) | 28 (55) | 21 (39)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 24 (44) | 24 (66)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 37 (80) | 32 (80)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes